CLINICAL TRIAL: NCT05097183
Title: Clinical Validation and Prognostic Evaluation of Accurate Commissural Alignment During Transcatheter Aortic Valve Implantation
Brief Title: Validation of Accurate Commissural Alignment During Transcatheter Aortic Valve Implantation
Acronym: ACA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ignacio J. Amat Santos (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Gerencia Regional de Salud de Castilla y Leon (Other)
Responsible Party: Sponsor-Investigator, Ignacio J. Amat Santos, Coordinator of Interventional Cardiology Unit, Hospital Clínico Universitario de Valladolid
Organization: Hospital Clínico Universitario de Valladolid (Other)
Other Study IDs: ICICOR-ACA-2021
Record Dates: First submitted 2021-10-15; First posted 2021-10-28 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Severe Aortic Valve Stenosis
Keywords: Transcatheter aortic valve replacement (TAVR)
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Transcatheter aortic valve replacement (TAVR) with standard procedure
- ACA: Transcatheter aortic valve replacement (TAVR) with Accurate Commissural Alignment (ACA) technique
  Interventions: Procedure: Accurate Commissural Alignment (ACA)

INTERVENTIONS:
Procedure: Accurate Commissural Alignment (ACA) — Software based, computed tomography analysis that allows planification of accurate commissural alignment of TAVR by inserting the delivery system in a patient-specific degree of rotation.
  Groups: ACA

SUMMARY:
Background: Transcatheter aortic valve replacement (TAVR) has become the preferred therapy for aortic stenosis. Given the growing life-expectancy, the risk of requiring coronary interventions or of developing prosthesis degeneration that could require TAVR-in-TAVR for its treatment progressively increases. During standard TAVI procedures the native and the prosthesis commissures are randomly aligned with misalignment in up to 70% of the cases. This might hinder coronary re-access in 18% of the cases, increase the risk of coronary obstruction during future TAVR-in-TAVR procedures, and has been associated to greater residual gradients.

Methods: Although several techniques have been developed to increase the degree of commissural alignment, all are imperfect or imply manipulation of the system within the patient, potentially increasing the risk of complications. The research team developed a software based on computed tomography analysis that allows planification of accurate commissural alignment by inserting the delivery system in a patient-specific degree of rotation.

Aim: The proponent team aimed to prospectively validate this methodology comparing a cohort of patients harboring TAVR with Acurate Commissural Alignment (ACA) vs. a control cohort with non-ACA standard technique, in order to determine benefits in terms of coronary re-access and clinical events (coronary events, valve degeneration, and TAVR-in-TAVR).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with severe aortic stenosis admitted to TAVR by Heart Team
* Pre-procedure CT-Scan for planning available.
* Signed informed consent.

Exclusion Criteria:

* Allergic to contrast
* Severe renal failure (GFR < 30 mL/min)
* Indication for chronic anticoagulation
* Horizontal aorta and/or severe aortic tortuosity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with severe aortic stenosis admitted to TAVR by Heart Team and fulfilling inclusion criteria in 16 centers in Spain. The Sponsor is proctoring the new ACA technique in this centers. TAVR patients treated both with standard and ACA technique will be included in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 274 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Degree of commissural alignment | 6 months
  Mean minimum angular deviation between TAVR posts and aortic valve commissures measured in CT-scan
Successful coronary re-access | 10 minutes, right after TAVR
  Coronary re-access was successful or not after TAVR implant
Presence of leaflet thrombosis | 6 months
  Presence of clinical/subclinical leaflets thrombosis assessed by CT-Scan

SECONDARY OUTCOMES:
Residual transvalvular gradients | 24 months
  Residual transvalvular gradients measured in transthoracic echocardiography

CONTACTS AND LOCATIONS:
Locations (15):
- Spain (15):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Clinic, Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitari Bellvitge, L'Hospitalet de Llobregat
  - Hospital clínico San Carlos, Madrid
  - Hospital La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital Virgen del Rocío, Seville
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Redondo A, Valencia-Serrano F, Santos-Martinez S, Delgado-Arana JR, Barrero A, Serrador A, Gutierrez H, Sanchez-Lite I, Sevilla T, Revilla A, Baladron C, Kim WK, Carrasco-Moraleja M, San Roman JA, Amat-Santos IJ. Accurate commissural alignment during ACURATE neo TAVI procedure. Proof of concept. Rev Esp Cardiol (Engl Ed). 2022 Mar;75(3):203-212. doi: 10.1016/j.rec.2021.02.004. Epub 2021 Mar 26. English, Spanish. PMID 33781722
- [Background] Redondo A, Santos-Martinez S, Delgado-Arana R, Baladron Zorita C, San Roman JA, Amat-Santos IJ. Fluoroscopic-based algorithm for commissural alignment assessment after transcatheter aortic valve implantation. Rev Esp Cardiol (Engl Ed). 2022 Feb;75(2):184-187. doi: 10.1016/j.rec.2021.08.010. Epub 2021 Sep 30. No abstract available. English, Spanish. PMID 34600863
- [Derived] Amat-Santos IJ, Gomez-Herrero J, Pinon P, Nombela-Franco L, Moreno R, Munoz-Garcia AJ, Redondo A, Gomez-Menchero A, Gomez-Salvador I, San Roman JA. Impact of commissural alignment on the hemodynamic performance of supra-annular self-expandable transcatheter aortic valves. Catheter Cardiovasc Interv. 2024 Nov;104(5):1060-1070. doi: 10.1002/ccd.31201. Epub 2024 Sep 10. PMID 39252591